## Effective Screening for Pain Study NCT01816763 July 2018

## Analysis plan

- 1. Describe study eligibility and enrollment.
  - Report numbers of patients approached, eligible/ineligible (reasons), enrolled/not enrolled (reasons), and analyzed/not analyzed in standard CONSORT figure (Figure 1)
  - b. Describe characteristics of study sample (numbers, percents, means) by randomized arm (Table 1)
- 2. Compare study measures
  - a. Describe results of Nurse NRS, NRS-one week assessed via table, PEG, (Table 2):
    - i. Mean (SD) score
    - ii. Percent of scores in no pain (0), mild (1-3), moderate (4-6), and severe (7+) categories.
  - b. Describe agreement on categories of pain severity: weighted kappa statistic for agreement of each screening measure compared with GCPS characteristic pain severity. (Table 3)

## Measure scoring

- 1) Calculate a score for each measure (all 0-10)
  - a) <u>Graded Chronic Pain Scale (GCPS) Characteristic Pain Intensity</u>: Sum of Pain Right Now (Q2) + Worst Pain (Q3) + Usual Pain Intensity (Q4)
    - i) Calculate score as above and divide by 3.
  - b) PEG: Sum 3 items and divide by 3.
  - c) NRS one-week
  - d) NRS nurse
- 2) For all measures, scores are rounded to the nearest whole number and categorized as follows:
  - a) No pain = 0
  - b) Mild pain = 1-3
  - c) Moderate pain = 4-6
  - d) Severe pain ≥ 7

## **Table 1: Characteristics of randomized participants**

| | Arm 1<br>(nurse NRS)<br>n= | Arm 2<br>(tablet NRS<br>average) n= | Arm 3 (PEG)<br>n= |
|---|---|---|---|
| Age, mean (SD) years | | | |
| Sex, n (%) male | | | |
| Race/ethnicity, n (%) | | | |
| White | | | |
| Black/African-American | | | |
| Asian | | | |
| Native American/Alaskan | | | |
| Native | | | |
| Native Hawaiian/Pacific | | | |
| Islander | | | |
| Hispanic/Latino | | | |

| Medical comorbidity score, |
|----------------------------|
| Seattle mean (SD) |
| Physical activity item |
| Friysical activity item |
| Disability days it an |
| Disability days item |
| Depression = (0/) (206.0) |
| Depression, n(%) (296.2x, |
| 296.3x, 300.4, 311) |
| Anxiety, n(%) (300.0x, |
| 300.2x) |
| PTSD, n(%) (309.81) |
| Alcohol use disorder, n(%) |
| (303.9x, 305.0x) |
| Drug use disorder, n(%) |
| (304.xx, 305.2x-305.7x, |
| 305.9x) |
| Back pain (codes TBD) |
| , , , |
| Joint pain (codes TBD) |
| , , |
| Headache (codes TBD) |
| , , , |
| Neuropathic pain (codes |
| TBD) |
| - |

Table 2: Pain screening outcomes by randomized arm

| | Arm 1<br>(usual<br>NRS)<br>n= | Arm 2<br>(tablet NRS<br>average)<br>n= | Arm 3<br>(PEG) n= | p-value |
|---|---|---|---|---|
| Screening measure score, mean (SD) | | | | |
| No pain (0), n (%) | | | | |
| Mild pain (1-3), n (%) | | | | |
| Moderate pain (4-6), n (%) | | | | |
| Severe pain (7+), n (%) | | | | |

Table 3: Agreement of screening measures with reference standard (GCPS characteristic pain intensity) on category of pain severity (none, mild, moderate, or severe)

| | None | Mild | Mod | Severe |
|--------------------|------|------|-----|--------|
| Usual NRS | | | | |
| Tablet NRS average | | | | |

| PEG |
|-----|